CLINICAL TRIAL: NCT02430194
Title: An Open-label, Dose-ranging, Proof-of-Concept Study to Evaluate the Safety and Efficacy of Lonafarnib With Ritonavir-Boosting +/- Peginterferon Alfa-2a in Patients Chronically Infected With Delta Hepatitis (HDV) (LOWR-2)
Brief Title: Lonafarnib Boosted With Ritonavir With and Without Peginterferon Alfa-2a (PEG IFN-a) in HDV (LOWR-2)
Acronym: LOWR-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eiger BioPharmaceuticals (Industry)
Collaborators: Ankara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EIG-300-Amendment 3
Expanded Access: NCT03895528 (Approved for marketing)
Record Dates: First submitted 2015-04-21; First posted 2015-04-30 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Chronic Hepatitis D Infection
MeSH Terms: interventions — lonafarnib; Ritonavir; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- lonafarnib/ritonavir - I (Experimental): lonafarnib 100 mg BID + ritonavir 100 mg QD
  Interventions: Drug: lonafarnib; Drug: ritonavir
- lonafarnib/ritonavir - II (Experimental): lonafarnib 100 mg BID + ritonavir 50 mg BID
  Interventions: Drug: lonafarnib; Drug: ritonavir
- lonafarnib/ritonavir - III (Experimental): lonafarnib 100 mg QD + ritonavir 100 mg QD
  Interventions: Drug: lonafarnib; Drug: ritonavir
- lonafarnib/ritonavir - IV (Experimental): lonafarnib 150 mg QD + ritonavir 100 mg QD
  Interventions: Drug: lonafarnib; Drug: ritonavir
- lonafarnib/ritonavir/PEG IFN-a - V (Experimental): lonafarnib 75 mg BID + ritonavir 100 mg BID (+ PEG IFN-a 180 ug QW on Week 12)
  Interventions: Drug: lonafarnib; Drug: ritonavir; Drug: Pegylated interferon-alfa-2a
- lonafarnib/ritonavir - VI (Experimental): lonafarnib 25 mg BID + ritonavir 100 mg BID
  Interventions: Drug: lonafarnib; Drug: ritonavir
- lonafarnib/ritonavir - VII (Experimental): lonafarnib 50 mg BID + ritonavir 100 mg BID
  Interventions: Drug: lonafarnib; Drug: ritonavir
- lonafarnib/ritonavir/PEG IFN-a - VIII (Experimental): lonafarnib 50 mg BID + ritonavir 100 mg BID (+ PEG IFN-a 180 ug QW on Week 12)
  Interventions: Drug: lonafarnib; Drug: ritonavir; Drug: Pegylated interferon-alfa-2a
- lonafarnib/ritonavir/PEG IFN-a - IX (Experimental): lonafarnib 25 mg BID + ritonavir 100 mg BID + PEG IFN-a 180 ug QW
  Interventions: Drug: lonafarnib; Drug: ritonavir; Drug: Pegylated interferon-alfa-2a
- lonafarnib/ritonavir/PEG IFN-a - X (Experimental): lonafarnib 50 mg BID + ritonavir 100 mg BID + PEG IFN-a 180 ug QW
  Interventions: Drug: lonafarnib; Drug: ritonavir; Drug: Pegylated interferon-alfa-2a

INTERVENTIONS:
Drug: lonafarnib — antiviral farnesyl transferase inhibitor
  Other Names: Sarasar, EBP994, LNF
Drug: ritonavir — CYP 3A4 inhibitor, lonafarnib booster
  Other Names: Norvir, RTV
Drug: Pegylated interferon-alfa-2a — immunomodulator
  Other Names: Pegasys; PEG IFN-alfa-2a; Peginterferon alfa-2a; PEG IFN-a
  Arms: lonafarnib/ritonavir/PEG IFN-a - IX; lonafarnib/ritonavir/PEG IFN-a - V; lonafarnib/ritonavir/PEG IFN-a - VIII; lonafarnib/ritonavir/PEG IFN-a - X

SUMMARY:
An Open-label, Dose-ranging Study to Evaluate the Safety and Efficacy of Lonafarnib with Ritonavir Boosting +/- Peginterferon alfa-2a in Patients Chronically Infected with Delta Hepatitis (HDV) (LOWR-2).

DETAILED DESCRIPTION:
Chronic delta hepatitis is a serious form of chronic liver disease caused by infection with the hepatitis D virus (HDV), a small RNA virus that requires farnesylation of its major structural protein (HDV antigen) for replication. Up to sixty subjects with chronic delta hepatitis will be randomized to receive one of ten different doses of lonafarnib. Dosing will occur over 12-48 weeks, and during that time, evidence of antiviral response will be assessed by frequent measurements of HDV-RNA. The primary therapeutic endpoint will be an improvement in quantitative serum HDV RNA levels after treatment with lonafarnib therapy. The primary safety endpoint will be the ability to tolerate the drug at the prescribed dose for the treatment duration. Several secondary endpoints will be measured, including side effects, ALT levels, and symptoms. Therapy will be stopped for intolerance to lonafarnib. This study is designed as a Phase 2a study assessing the safety, tolerance and antiviral activity of nine dosing combinations of lonafarnib with ritonavir boosting with and without peginterferon alfa-2a (PEG IFN-a).

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 18 to 65 years of age who are diagnosed with HDV by PCR
* Chronic hepatitis D infection, genotype 1, documented by a positive anti-HDV Ab test at least of 6 months duration and detectable HDV RNA by PCR within 3 months to study entry
* Liver biopsy within the last two years (biopsy can be done at the Screening Visit)
* Positive viral load of >100,000 copies/mL as measured by quantitative PCR
* Electrocardiogram (ECG) shows no acute ischemia or clinically significant abnormality and a QT/QTc interval <450 milliseconds - using Bazett's correction
* Females of childbearing potential (intact uterus and within 1 year since the last menstrual period) should be non-lactating and have a negative serum pregnancy test. In addition, these subjects should agree to use one of the following acceptable birth control methods throughout the study:

  1. abstinence
  2. surgical sterilization (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) six months minimum
  3. IUD in place for at least six months
  4. barrier methods (condom or diaphragm) with spermicide
  5. surgical sterilization of the partner (vasectomy for six months)
  6. hormonal contraceptives for at least three months prior to the first dose of study drug
* Willing and able to comply with study procedures and provide written informed consent

Exclusion Criteria:

* Participation in a clinical trial with or use of any investigational agent within 30 days of Study Visit 1
* Patients co-infected with HIV
* Patients with screening tests positive for HCV, or anti-HIV Ab
* History of decompensated cirrhosis within the past year
* Active jaundice defined by total bilirubin > 2.0 excluding Gilbert's disease
* INR ≥ 1.5
* Eating disorder or alcohol abuse within the past 2 years, excessive alcohol intake (> 20 g per day for females (1.5 standard alcohol drinks) or > 30 g per day for males (2.0 standard alcohol drinks) (a standard drink contains 14 g of alcohol: 12 oz of beer, 5 oz of wine or 1.5 oz of spirits) (1.0 fluid oz (US) = 29.57 mL)
* Drug abuse within the last six months with the exception of cannabinoids and their derivatives
* Patients with absolute neutrophil count (ANC) < 1500 cells/mm^3; platelet count < 100,000 cells/mm^3; hemoglobin < 12 g/dL for women and < 13 g/dL for men; abnormal TSH,T4, or T3 or thyroid function not adequately controlled; or serum creatinine concentration ≥ 1.5 times upper limit of normal (ULN)
* History or clinical evidence of any of the following:

  1. variceal bleeding, ascites, hepatic encephalopathy, CTP score > 6, decompensated liver disease or any other form of non-viral hepatitis
  2. immunologically mediated disease (e.g., rheumatoid arthritis, inflammatory bowel disease, severe psoriasis, systemic lupus erythematosus) requiring more than intermittent nonsteroidal anti-inflammatory medications for management or that requires frequent or prolonged use of corticosteroids (inhaled asthma medications are allowed)
  3. any malignancy within 3 years except for basal cell skin cancer
  4. significant or unstable cardiac disease (e.g., angina, congestive heart failure, uncontrolled hypertension, history of arrhythmia)
  5. chronic pulmonary disease (e.g., chronic obstructive pulmonary disease) associated with functional impairment
  6. severe or uncontrolled psychiatric disease, including severe depression, history of suicidal ideation, suicidal attempts or psychosis requiring medication and/or hospitalization 2
* Patients with a body mass index > 30 kg/m^2
* Concomitant drugs known to prolong the QT interval

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cihan Yurdaydin, MD, Principal Investigator — Ankara University
Locations (1):
- Ankara University Medical School, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yurdaydin C, Keskin O, Yurdcu E, Caliskan A, Onem S, Karakaya F, Kalkan C, Karatayli E, Karatayli S, Choong I, Apelian D, Koh C, Heller T, Idilman R, Bozdayi AM, Glenn JS. A phase 2 dose-finding study of lonafarnib and ritonavir with or without interferon alpha for chronic delta hepatitis. Hepatology. 2022 Jun;75(6):1551-1565. doi: 10.1002/hep.32259. Epub 2021 Dec 23. PMID 34860418
- See also: Eiger BioPharmaceuticals company website — http://eigerbio.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Lonafarnib/Ritonavir/PEG IFN-alfa-2a - V: lonafarnib 75 mg BID + ritonavir 100 mg BID; + PEG IFN-alfa-2a 180 ug QW on Week 12
  lonafarnib: antiviral farnesyl transferase inhibitor
  ritonavir: CYP 3A4 inhibitor, lonafarnib booster
  PEG IFN-alfa-2a: immunomodulator
- Lonafarnib/Ritonavir/PEG IFN-alfa-2a - VII: lonafarnib 50 mg BID + ritonavir 100 mg BID; + PEG IFN-alfa-2a 180 ug QW;
  lonafarnib: antiviral farnesyl transferase inhibitor
  ritonavir: CYP 3A4 inhibitor, lonafarnib booster
  PEG IFN-alfa-2a: immunomodulator
- Lonafarnib/Ritonavir/PEG IFN-alfa-2a - VIII: lonafarnib 50 mg BID + ritonavir 100 mg BID; + PEG IFN-alfa-2a 180 ug QW on Week 12
  lonafarnib: antiviral farnesyl transferase inhibitor
  ritonavir: CYP 3A4 inhibitor, lonafarnib booster
  PEG IFN-alfa-2a: immunomodulator
- Lonafarnib/Ritonavir - IX: lonafarnib 50 mg BID + ritonavir 100 mg BID
  lonafarnib: antiviral farnesyl transferase inhibitor
  ritonavir: CYP 3A4 inhibitor, lonafarnib booster
- Lonafarnib/Ritonavir/PEG IFN-alfa-2a - X: lonafarnib 25 mg BID + ritonavir 100 mg BID + PEG IFN-alfa-2a 180 ug QW
  lonafarnib: antiviral farnesyl transferase inhibitor
  ritonavir: CYP 3A4 inhibitor, lonafarnib booster
  PEG IFN-alfa-2a: immunomodulator
Period: Overall Study
Arm/Group | Lonafarnib/Ritonavir - I | Lonafarnib/Ritonavir - II | Lonafarnib/Ritonavir - III | Lonafarnib/Ritonavir - IV | Lonafarnib/Ritonavir/PEG IFN-alfa-2a - V | Lonafarnib/Ritonavir - VI | Lonafarnib/Ritonavir/PEG IFN-alfa-2a - VII | Lonafarnib/Ritonavir/PEG IFN-alfa-2a - VIII | Lonafarnib/Ritonavir - IX | Lonafarnib/Ritonavir/PEG IFN-alfa-2a - X
Started | 4 | 4 | 5 | 3 | 3 | 6 | 13 | 5 | 7 | 5
Completed | 3 | 3 | 3 | 3 | 3 | 6 | 11 | 4 | 3 | 5
Not Completed | 1 | 1 | 2 | 0 | 0 | 0 | 2 | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Population: 18-year-old to 65-year-old patients with chronic HDV infection, documented by a positive anti-HDV test of at least 6 month duration and detectable HDV RNA by PCR within 3 months to study entry, were included. All patients were required to be HDV RNA-positive at baseline and have compensated liver disease. Platelet and white blood cell counts had to be ≥100,000 (×10^9/L) and 3000 (×10^9/L), respectively.
Groups:
- Lonafarnib/Ritonavir - V: lonafarnib 75 mg BID + ritonavir 100 mg BID + PEG IFN-a 180 ug QW on Week 12
  lonafarnib: antiviral farnesyl transferase inhibitor
  Ritonavir: CYP 3A4 inhibitor, lonafarnib booster
  PEG IFN-a: immunomodulator
- Lonafarnib/Ritonavir/PEG IFN-a - VIII: lonafarnib 50 mg BID + ritonavir 100 mg BID + PEG IFN-a 180 ug QW on Week 12
  lonafarnib: antiviral farnesyl transferase inhibitor
  Ritonavir: CYP 3A4 inhibitor, lonafarnib booster
  PEG IFN-a: immunomodulator
- Lonafarnib/Ritonavir/PEG IFN-a - IX: lonafarnib 50 mg BID + ritonavir 100 mg BID + PEG IFN-a 180 ug QW
  lonafarnib: antiviral farnesyl transferase inhibitor
  Ritonavir: CYP 3A4 inhibitor, lonafarnib booster
  PEG IFN-a: immunomodulator
- Lonafarnib/Ritonavir - X: lonafarnib 25 mg BID + ritonavir 100 mg BID + PEG IFN-a 180 ug QW
  lonafarnib: antiviral farnesyl transferase inhibitor
  Ritonavir: CYP 3A4 inhibitor, lonafarnib booster
  PEG IFN-a: immunomodulator
- Total: Total of all reporting groups
Arm/Group | Lonafarnib/Ritonavir - I | Lonafarnib/Ritonavir - II | Lonafarnib/Ritonavir - III | Lonafarnib/Ritonavir - IV | Lonafarnib/Ritonavir - V | Lonafarnib/Ritonavir - VI | Lonafarnib/Ritonavir - VII | Lonafarnib/Ritonavir/PEG IFN-a - VIII | Lonafarnib/Ritonavir/PEG IFN-a - IX | Lonafarnib/Ritonavir - X | Total
Number analyzed (Participants) | 4 | 4 | 5 | 3 | 3 | 6 | 13 | 5 | 7 | 5 | 55
Age, Continuous [Median (Full Range); unit: years] — 3 enrolled subjects were above the age limit for eligibility: 1 subject in the lonafarnib/ritonavir - III group and 2 subjects in the lonafarnib/ritonavir - VII group.
  years | 31 [23 to 40] | 51 [37 to 54] | 61 [53 to 66] | 56 [42 to 60] | 59 [58 to 61] | 49 [31 to 57] | 41 [27 to 70] | 39 [25 to 52] | 50 [41 to 59] | 39 [29 to 58] | 50 [23 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 3 | 0 | 1 | 3 | 6 | 0 | 4 | 2 | 19
  Male | 4 | 4 | 2 | 3 | 2 | 3 | 7 | 5 | 3 | 3 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 4 | 5 | 3 | 3 | 6 | 13 | 5 | 7 | 5 | 55
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 4 | 4 | 5 | 3 | 3 | 6 | 13 | 5 | 7 | 5 | 55

OUTCOME MEASURES:

1. Primary Outcome: ≥2 log10 Decline of HDV RNA From Baseline at End of Treatment (EOT)
Description: Proportion of intent to treat patients with ≥2 log10 decline of HDV RNA from baseline at end of treatment (EOT)
Time Frame: 12-48 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Lonafarnib/Ritonavir - I: lonafarnib 100 mg BID + ritonavir 100 mg QD for 12 weeks
- Lonafarnib/Ritonavir - II: lonafarnib 100 mg BID + ritonavir 50 mg BID for 12 weeks
- Lonafarnib/Ritonavir - III: lonafarnib 100 mg QD + ritonavir 100 mg QD for 12 weeks
- Lonafarnib/Ritonavir - IV: lonafarnib 150 mg QD + ritonavir 100 mg QD for 12 weeks
- Lonafarnib/Ritonavir/PEG IFN-a - V: lonafarnib 75 mg BID + ritonavir 100 mg BID for 12 weeks; + PEG IFN-a 180 ug QW on Week 12-24
- Lonafarnib/Ritonavir - VI: lonafarnib 25 mg BID + ritonavir 100 mg BID for 24 weeks
- Lonafarnib/Ritonavir - VII: lonafarnib 50 mg BID + ritonavir 100 mg BID for 24 weeks
- Lonafarnib/Ritonavir/PEG IFN-a - VIII: lonafarnib 50 mg BID + ritonavir 100 mg BID for 12 weeks; + PEG IFN-a 180 ug QW on Week 12-24
- Lonafarnib/Ritonavir/PEG IFN-a - IX: lonafarnib 25 mg BID + ritonavir 100 mg BID + PEG IFN-a 180 ug QW for 24 weeks
- Lonafarnib/Ritonavir/PEG IFN-a - X: lonafarnib 50 mg BID + ritonavir 100 mg BID + PEG IFN-a 180 ug QW for 24 weeks
Arm/Group | Lonafarnib/Ritonavir - I | Lonafarnib/Ritonavir - II | Lonafarnib/Ritonavir - III | Lonafarnib/Ritonavir - IV | Lonafarnib/Ritonavir/PEG IFN-a - V | Lonafarnib/Ritonavir - VI | Lonafarnib/Ritonavir - VII | Lonafarnib/Ritonavir/PEG IFN-a - VIII | Lonafarnib/Ritonavir/PEG IFN-a - IX | Lonafarnib/Ritonavir/PEG IFN-a - X
Number analyzed (Participants) | 4 | 4 | 5 | 3 | 3 | 6 | 13 | 5 | 7 | 5
Participants | 1 | 0 | 1 | 0 | 1 | 1 | 5 | 4 | 3 | 4

2. Secondary Outcome: < LLOQ in HDV RNA at End of Treatment (EOT)
Description: Proportion of intent to treat patients with HDV RNA below the limit of quantitation at end of treatment
Time Frame: 12-48 weeks
Population: intent to treat population
Measure: Count of Participants; unit: Participants
Groups:
- Lonafarnib/Ritonavir/PEG IFN-a - V: lonafarnib 75 mg BID + ritonavir 100 mg BID for 12 weeks; + PEG IFNa 180 mcg QW from Week 12-24
- Lonafarnib/Ritonavir/PEG IFN-a - VIII: lonafarnib 50 mg BID + ritonavir 100 mg BID for 12 weeks; + PEG IFN-a 180 ug QW from Week 12-24
- Lonafarnib/Ritonavir/PEG IFN-a - IX: lonafarnib 25 mg BID + ritonavir 100 mg BID + PEG IFN-a 180 mcg QW for 24 weeks
- Lonafarnib/Ritonavir/PEG IFN-a - X: lonafarnib 50 mg BID + ritonavir 100 mg BID + PEG IFN-a 180 mcg QW for 24 weeks
Arm/Group | Lonafarnib/Ritonavir - I | Lonafarnib/Ritonavir - II | Lonafarnib/Ritonavir - III | Lonafarnib/Ritonavir - IV | Lonafarnib/Ritonavir/PEG IFN-a - V | Lonafarnib/Ritonavir - VI | Lonafarnib/Ritonavir - VII | Lonafarnib/Ritonavir/PEG IFN-a - VIII | Lonafarnib/Ritonavir/PEG IFN-a - IX | Lonafarnib/Ritonavir/PEG IFN-a - X
Number analyzed (Participants) | 4 | 4 | 5 | 3 | 3 | 6 | 13 | 5 | 7 | 5
Participants | 0 | 1 | 1 | 0 | 1 | 0 | 6 | 1 | 3 | 2

3. Secondary Outcome: ALT Normalization at End of Treatment
Description: Proportion of intent to treat population who normalize ALT at end of treatment
Time Frame: 12-48 weeks
Population: intent to treat population
Measure: Count of Participants; unit: Participants
Groups:
- Lonafarnib/Ritonavir - V: lonafarnib 75 mg BID + ritonavir 100 mg BID for 12 weeks; + PEG IFN-a 180 mcg QW from Week 12-24
- Lonafarnib/Ritonavir - VI: lonafarnib 25 mg BID + ritonavir 100 mg BID for 12 weeks
- Lonafarnib/Ritonavir - VII: lonafarnib 50 mg BID + ritonavir 100 mg BID for 12 weeks
- Lonafarnib/Ritonavir/PEG IFN-a - VIII: lonafarnib 50 mg BID + ritonavir 100 mg BID for 12 weeks; + PEG IFN-a 180 mcg QW from Week 12-24
- Lonafarnib/Ritonavir/PEG IFN-a - X: lonafarnib 25 mg BID + ritonavir 100 mg BID + PEG IFN-a 180 mcg QW for 24 weeks
Arm/Group | Lonafarnib/Ritonavir - I | Lonafarnib/Ritonavir - II | Lonafarnib/Ritonavir - III | Lonafarnib/Ritonavir - IV | Lonafarnib/Ritonavir - V | Lonafarnib/Ritonavir - VI | Lonafarnib/Ritonavir - VII | Lonafarnib/Ritonavir/PEG IFN-a - VIII | Lonafarnib/Ritonavir/PEG IFN-a - IX | Lonafarnib/Ritonavir/PEG IFN-a - X
Number analyzed (Participants) | 4 | 4 | 5 | 3 | 3 | 6 | 13 | 5 | 7 | 5
Participants | 3 | 1 | 1 | 2 | 0 | 2 | 6 | 0 | 5 | 2

4. Other Pre Specified Outcome: Mean HDV RNA Decline
Description: mean HDV RNA decline of intent to treat population from baseline to end of treatment
Time Frame: 12-48 weeks
Population: intent to treat population
Measure: Mean (Standard Error); unit: log HDV RNA IU/mL
Groups:
- Lonafarnib/Ritonavir/PEG IFN-a - V: lonafarnib 75 mg BID + ritonavir 100 mg BID; + PEG IFN-a 180 ug QW from Week 12-24
- Lonafarnib/Ritonavir/PEG IFN-a - VIII: lonafarnib 50 mg BID + ritonavir 100 mg BID; + PEG IFN-a 180 ug QW from Week 12-24
Arm/Group | Lonafarnib/Ritonavir - I | Lonafarnib/Ritonavir - II | Lonafarnib/Ritonavir - III | Lonafarnib/Ritonavir - IV | Lonafarnib/Ritonavir/PEG IFN-a - V | Lonafarnib/Ritonavir - VI | Lonafarnib/Ritonavir - VII | Lonafarnib/Ritonavir/PEG IFN-a - VIII | Lonafarnib/Ritonavir/PEG IFN-a - IX | Lonafarnib/Ritonavir/PEG IFN-a - X
Number analyzed (Participants) | 4 | 4 | 5 | 3 | 3 | 6 | 13 | 5 | 7 | 5
log HDV RNA IU/mL | -1.39 (1.27) | 0.33 (1.08) | -1.11 (3.1) | -0.67 (0.24) | -1.97 (1.6) | -0.31 (1.61) | -1.94 (1.3) | -2.85 (0.49) | -2.69 (1.66) | -3.81 (0.94)

ADVERSE EVENTS:
Time Frame: treatment period 12-48 weeks
Arm/Group | Lonafarnib/Ritonavir - I | Lonafarnib/Ritonavir - II | Lonafarnib/Ritonavir - III | Lonafarnib/Ritonavir - IV | Lonafarnib/Ritonavir/PEG IFN-a - V | Lonafarnib/Ritonavir - VI | Lonafarnib/Ritonavir - VII | Lonafarnib/Ritonavir/PEG IFN-a - VIII | Lonafarnib/Ritonavir/PEG IFN-a - IX | Lonafarnib/Ritonavir/PEG IFN-a - X
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/5 | 0/3 | 0/3 | 0/6 | 0/13 | 0/5 | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 3/5 | 0/3 | 0/3 | 0/6 | 2/13 | 1/5 | 1/7 | 1/5
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 5/5 | 3/3 | 3/3 | 6/6 | 13/13 | 5/5 | 7/7 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lonafarnib/Ritonavir - I (N=4) | Lonafarnib/Ritonavir - II (N=4) | Lonafarnib/Ritonavir - III (N=5) | Lonafarnib/Ritonavir - IV (N=3) | Lonafarnib/Ritonavir/PEG IFN-a - V (N=3) | Lonafarnib/Ritonavir - VI (N=6) | Lonafarnib/Ritonavir - VII (N=13) | Lonafarnib/Ritonavir/PEG IFN-a - VIII (N=5) | Lonafarnib/Ritonavir/PEG IFN-a - IX (N=7) | Lonafarnib/Ritonavir/PEG IFN-a - X (N=5)
diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
fatigue (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
hepatic decompensation (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
neuropathy vasculitis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lonafarnib/Ritonavir - I (N=4) | Lonafarnib/Ritonavir - II (N=4) | Lonafarnib/Ritonavir - III (N=5) | Lonafarnib/Ritonavir - IV (N=3) | Lonafarnib/Ritonavir/PEG IFN-a - V (N=3) | Lonafarnib/Ritonavir - VI (N=6) | Lonafarnib/Ritonavir - VII (N=13) | Lonafarnib/Ritonavir/PEG IFN-a - VIII (N=5) | Lonafarnib/Ritonavir/PEG IFN-a - IX (N=7) | Lonafarnib/Ritonavir/PEG IFN-a - X (N=5)
diarrhea (Gastrointestinal disorders) | 3 | 2 | 3 | 2 | 3 | 3 | 9 | 5 | 3 | 5
nausea (Gastrointestinal disorders) | 2 | 2 | 3 | 2 | 3 | 4 | 8 | 4 | 4 | 3
vomiting (Gastrointestinal disorders) | 0 | 1 | 3 | 1 | 0 | 2 | 7 | 1 | 1 | 1
fatigue (General disorders) | 3 | 3 | 4 | 3 | 3 | 4 | 10 | 5 | 4 | 5
anorexia (Gastrointestinal disorders) | 3 | 4 | 2 | 3 | 3 | 2 | 8 | 4 | 2 | 4
weight loss (Investigations) | 3 | 2 | 2 | 3 | 2 | 3 | 7 | 3 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-10): https://cdn.clinicaltrials.gov/large-docs/94/NCT02430194/Prot_SAP_000.pdf